CLINICAL TRIAL: NCT03977376
Title: Effectiveness of a Prequirurgic Instrument to Decrease Anxiety in Urogical Quirurgic Patients: a Randomized Clinical Trial
Acronym: EPECA30-2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Carmen Gracia Ruiz García, Máster Social-sanitary Science Investigation, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPECA30-2018
Record Dates: First submitted 2019-06-02; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Anxiety; Nurse-Patient Relations; Behavior
Keywords: anxiety; Urogical; Guide of Hosting; Comunication instrument; Patients
MeSH Terms: conditions — Anxiety Disorders; Behavior

STUDY DESIGN:
Masking Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Valuation instruments were two validated scales: ESAS y HADS. Experimental nursing instrument: Guide of hosting.
  Interventions: Other: Guide of hosting
- Control (No Intervention): Valuation instruments were two validated scales: ESAS y HADS. Without Guide of hosting.

INTERVENTIONS:
Other: Guide of hosting — Guide of hosting with information about hospitalization to decrease anxiety
  Arms: Intervention

SUMMARY:
The overall aim of this program of research is to decrease anxiety in urogical scheduled patients for surgical intervention developing an nursing comunication instrument: a Guide of Hosting for urogical scheduled patients for surgical intervention.

DETAILED DESCRIPTION:
The overall aim of this program of research is to decrease anxiety in urogical scheduled patients for surgical intervention developing an nursing communication instrument: a Guide of Hosting for urological scheduled patients for surgical intervention.

The purpose of the proposed project is to establish the feasibility and acceptability of this guide to decrease the anxiety in this patients, using a randomized clinical trial like a research design, which would test the effectiveness of this communication instrument in comparation to a control condition (patients without guide of housting).

To achieve the investigators specific aims, the investigator conducted a randomized clinical trial (n=50), with two groups: intervention group (with Guide of Hosting) and control group (which shows a control condition).

Valuation instruments were two validated scales: ESAS y HADS. Anxiety was the primary outcome variable assessed in the RCT; depression and pain were a secondary outcomes variables.

ELIGIBILITY:
Inclusion Criteria:

* Age limits: 18 years old.
* with hospital admission scheduled at 5ªA hospitalization service of the University Hospital of Guadalajara for surgical intervention with urological diagnosis

Exclusion Criteria:

* patients with cognitive deficit.
* patients with recurrent insomnia problems
* without Spanish language proficiency
* patients that have participated in a clinical trial in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-26 (Actual)

PRIMARY OUTCOMES:
Anxiety: Hospital Anxiety and Depression Scale (HADS) | 4-5 months
  To assess anxiety and depressive symptoms in a general medical population. There are 7 depression items measuring cognitive and emotional aspects of depression, predominantly anhedonia, intermingled with 7 anxiety items that focus on cognitive and emotional aspects of anxiety. Somatic items relating to emotional and physical disorders are excluded.
  With 14 items.
Anxiety: Edmonton Symptom Assessment System (ESAS) | 4-5 months
  Value scale ESAS is a widely used, self-report symptom intensity tool for assessing nine common symptoms in hospilatation, with ratings ranging from 0 (none, best) to 10 (worst).

SECONDARY OUTCOMES:
Pain: Edmonton Symptom Assessment System (ESAS) | 4-5 months
  Value scale ESAS is a widely used, self-report symptom intensity tool for assessing nine common symptoms in hospitalitation, with ratings ranging from 0 (none, best) to 10 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gracia Ruiz Garcia, Principal Investigator — Máster Universitario en Investigación en Ciencias Sociosanitarias - UAH
Locations (1):
- EPECA, Guadalajara, Spain

IPD SHARING:
Plan to Share IPD: No